CLINICAL TRIAL: NCT03891082
Title: A Comparative Study Between Bakri Balloon and B Lynch Suture Used to Control Primary Postpartum Hemorrhage After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52
Record Dates: First submitted 2019-03-24; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-Lynch (Active Comparator): A 70 mm round bodied hand needle on which a No. 2 absorbable suture is mounted is used to puncture the uterus 3 cm from the right lower edge of the uterine incision and 3 cm from the right lateral border. The mounted No. 2 absorbable suture is threaded through the uterine cavity to emerge at the upper incision margin 3 cm above and approximately 4 cm from the lateral border.The absorbable suture is fed posteriorly and vertically to enter the posterior wall of the uterine cavity at the same level as the upper anterior entry point.
  Interventions: Procedure: B-Lynch
- Bakri balloon (Active Comparator): Insert the balloon portion of the catheter in the uterus; making certain that the entire balloon is inserted past the cervical canal and internal ostium.
  Interventions: Procedure: BALLOON INSERTION

INTERVENTIONS:
Procedure: B-Lynch — A 70 mm round bodied hand needle on which a No. 2 absorbable suture is mounted is used to puncture the uterus 3 cm from the right lower edge of the uterine incision and 3 cm from the right lateral border. The mounted No. 2 absorbable suture is threaded through the uterine cavity to emerge at the upper incision margin 3 cm above and approximately 4 cm from the lateral border
  Arms: B-Lynch
Procedure: BALLOON INSERTION — Insert the balloon portion of the catheter in the uterus; making certain that the entire balloon is inserted past the cervical canal and internal ostium. NOTE: Avoid excessive force when inserting the balloon into the uterus. Place a Foley catheter in patient bladder to collect and monitor urine output. To ensure maintenance of correct placement and maximize tamponade effect, the vaginal canal may be packed with iodine or antibiotic soaked vaginal gauze at this time.
  Other Names: Bakri balloon:
  Arms: Bakri balloon

SUMMARY:
Hundred (100) patients with primary postpartum hemorrhage during caesarean section due to atonic uterus will be recruited for this study.and randomized to either B lynch or Bakeri Ballon

B-Lynch:

A 70 mm round bodied hand needle on which a No. 2 absorbable suture is mounted is used to puncture the uterus 3 cm from the right lower edge of the uterine incision and 3 cm from the right lateral border. The mounted No. 2 absorbable suture is threaded through the uterine cavity to emerge at the upper incision margin 3 cm above and approximately 4 cm from the lateral border (because the uterus widens from below upwards). The absorbable suture now visible is passed over to compress the uterine fundus approximately 34 cm from the right cornual border. The absorbable suture is fed posteriorly and vertically to enter the posterior wall of the uterine cavity at the same level as the upper anterior entry point. The absorbable suture is pulled under moderate tension assisted by manual compression exerted by the first assistant. The length of the absorbable suture is passed back posteriorly through the same surface marking as for the right side, the suture lying horizontally. The absorbable suture is fed through posteriorly and vertically over the fundus to lie anteriorly and Research Template 7 Final Version: 1/6/2018 vertically compressing the fundus on the left side as occurred on the right. The needle is passed in the same fashion on the left side through the uterine cavity and out approximately 3 cm anteriorly and below the lower incision margin on the left side. The two lengths of absorbable suture are pulled taught assisted by bi-manual compression to minimize trauma and to achieve or aid compression. During such compression the vagina is checked that the bleeding is controlled. As good hemostasis is secured and whilst the uterus is compressed by an experienced assistant the principal surgeon throws a knot (double throw) followed by two or three further throws to secure tension. The lower transverse uterine incision is now closed in the normal way, in two layers, with or without closure of the lower uterine segment peritoneum. BALLOON INSERTION Insert the balloon portion of the catheter in the uterus; making certain that the entire balloon is inserted past the cervical canal and internal ostium. NOTE: Avoid excessive force when inserting the balloon into the uterus. Place a Foley catheter in patient bladder to collect and monitor urine output. To ensure maintenance of correct placement and maximize tamponade effect, the vaginal canal may be packed with iodine or antibiotic soaked vaginal gauze at this time.

DETAILED DESCRIPTION:
Hundred (100) patients with primary postpartum hemorrhage during caesarean section due to atonic uterus will be recruited for this study.and randomized to either B lynch or Bakeri Ballon

B-Lynch:

A 70 mm round bodied hand needle on which a No. 2 absorbable suture is mounted is used to puncture the uterus 3 cm from the right lower edge of the uterine incision and 3 cm from the right lateral border. The mounted No. 2 absorbable suture is threaded through the uterine cavity to emerge at the upper incision margin 3 cm above and approximately 4 cm from the lateral border (because the uterus widens from below upwards). The absorbable suture now visible is passed over to compress the uterine fundus approximately 34 cm from the right cornual border. The absorbable suture is fed posteriorly and vertically to enter the posterior wall of the uterine cavity at the same level as the upper anterior entry point. The absorbable suture is pulled under moderate tension assisted by manual compression exerted by the first assistant. The length of the absorbable suture is passed back posteriorly through the same surface marking as for the right side, the suture lying horizontally. The absorbable suture is fed through posteriorly and vertically over the fundus to lie anteriorly and Research Template 7 Final Version: 1/6/2018 vertically compressing the fundus on the left side as occurred on the right. The needle is passed in the same fashion on the left side through the uterine cavity and out approximately 3 cm anteriorly and below the lower incision margin on the left side. The two lengths of absorbable suture are pulled taught assisted by bi-manual compression to minimize trauma and to achieve or aid compression. During such compression the vagina is checked that the bleeding is controlled. As good hemostasis is secured and whilst the uterus is compressed by an experienced assistant the principal surgeon throws a knot (double throw) followed by two or three further throws to secure tension. The lower transverse uterine incision is now closed in the normal way, in two layers, with or without closure of the lower uterine segment peritoneum. BALLOON INSERTION Insert the balloon portion of the catheter in the uterus; making certain that the entire balloon is inserted past the cervical canal and internal ostium. NOTE: Avoid excessive force when inserting the balloon into the uterus. Place a Foley catheter in patient bladder to collect and monitor urine output. To ensure maintenance of correct placement and maximize tamponade effect, the vaginal canal may be packed with iodine or antibiotic soaked vaginal gauze at this time.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing caesarean sections landing up in atonic PPH during LSCS with failure of medical line of management:

  1. Full term pregnancy
  2. Didn't complete her family
  3. Elective caesarian section

Exclusion Criteria:

* 1.) PPH after vaginal delivery 2.) Secondary PPH 3.) PPH due to causes other than atonicity 4.) Antepartum hemorrhage cases 5.) Patients with bleeding tendency 6.) If any complication occurred during caesarian section (e.g. bladder injury, DIC)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Estimation of blood loss: | during the operation
  number of saturated pads + amount in suction container (if used) + visualization by the operating team.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Professor

REFERENCES:
- [Derived] Kellie FJ, Wandabwa JN, Mousa HA, Weeks AD. Mechanical and surgical interventions for treating primary postpartum haemorrhage. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013663. doi: 10.1002/14651858.CD013663. PMID 32609374